CLINICAL TRIAL: NCT00663845
Title: A Randomized, Double-blind, Placebo-controlled, Parallel-group, Study Evaluating the Efficacy, Safety, and Duration of Erection of Flexible-dose Vardenafil Administered for 12 Weeks Compared to Placebo in Subjects With Erectile Dysfunction and Dyslipidemia.
Brief Title: Assessing Efficacy and Safety of Flexible Dosing With Vardenafil in Subjects With Erectile Dysfunction and Hyperlipidemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12165
Record Dates: First submitted 2008-04-17; First posted 2008-04-22 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Erectile Dysfunction
Keywords: Male Erectile Dysfunction; Dyslipidemia; Vardenafil
MeSH Terms: conditions — Erectile Dysfunction; Dyslipidemias | interventions — Vardenafil Dihydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental)
  Interventions: Drug: Levitra (Vardenafil, BAY38-9456)
- Arm 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levitra (Vardenafil, BAY38-9456) — 10mg Vardenafil taken orally 1h prior to sexual intercourse
  Arms: Arm 1
Drug: Placebo — Matching placebo
  Arms: Arm 2

SUMMARY:
This study is being conducted in US to obtain information on the efficacy, safety, and duration of erection of flexible-dose regime of vardenafil compared to placebo (dummy medication with no pharmacological activity), in patients with co-morbid factors associated with erectile dysfunction (also called impotence). The duration of erection endpoint will be assessed by patient utilized stopwatch timings during each attempt at sexual intercourse. Elevated levels of total cholesterol or low levels of HDL may result in atherosclerosis and induce erectile dysfunction. Vardenafil (Levitra) is approved by the Food and Drug Administration for the treatment of erectile dysfunction. While there is no intent to assess the effect vardenafil has on blood lipids, the study will provide prospective data on men diagnosed with both ED and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

* Males with ED for more than 6 months, according to the NIH Consensus Statement (inability to attain and/or maintain penile erection sufficient for satisfactory sexual performance)
* Stable heterosexual relationship for more than 6 months
* Between 18 and <65 years of age
* Diagnosed dyslipidemia and treated with a stable dose of a statin (or generic equivalent) >/=3 months at Screening. In addition, the subject must have remained on this stable dose of statin (or its generic equivalent) throughout the study and no additional therapy to treat dyslipidemia was initiated
* InternationaI Index of Erectile Function - Erectile Function domain score of <25, denoting mild to severe ED at Visit 2

Exclusion Criteria:

* Primary hypoactive sexual desire
* History of myocardial infarction, stroke or life-threatening arrhythmia within prior 6 month
* Nitrate therapy
* Other exclusion criteria apply according to the US Product Information

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2006-05; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Sexual Encounter Profile Question 2 and 3 and International Index of Erectile Function - Erectile Function domain | 12 weeks

SECONDARY OUTCOMES:
Duration of erection leading to positive Sexual Encounter Profile Question 3 | 12 weeks
Safety and tolerability | 12 weeks
Other patient diary based variables | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer